CLINICAL TRIAL: NCT00047450
Title: Citalopram Augmentation in Older Patients With Schizophrenia
Brief Title: Antidepressant Treatment in Older Adults With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sidney Zisook, Research Scientist, Veterans Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH063931 (NIH); R01MH063931 (NIH); DATR A4-GPX; NCT00046098 (obsolete NCT alias)
Record Dates: First submitted 2002-10-04; First posted 2002-10-07 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Schizophrenia
Keywords: Psychotic Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Participants will take placebo
  Interventions: Drug: Placebo
- 2 (Active Comparator): Participants will take citalopram (Celexa)
  Interventions: Drug: Citalopram (Celexa)

INTERVENTIONS:
Drug: Citalopram (Celexa) — Citalopram for 3 months
  Arms: 2
Drug: Placebo — Placebo for 3 months
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of citalopram (Celexa) for the treatment of depressive symptoms in middle-aged and elderly patients with schizophrenia.

DETAILED DESCRIPTION:
Older people with schizophrenia suffer from greater physical comorbidity, cognitive impairment, and medication side effects compared to their younger counterparts. Unfortunately, little research is available to guide the treatment of subsyndromal depressive symptoms in older adults. This study will compare the antidepressant citalopram to placebo to determine the most effective treatment for reducing depressive symptoms in older patients with schizophrenia

After patients have been on stable treatment with antipsychotic medication for at least 4 weeks, they are randomly assigned to receive antipsychotic medication plus either citalopram or placebo for 3 months. Depressive symptoms and side effects are assessed weekly for the first month, biweekly for the second month, and again at the end of the third month. Cognition, motor and daily functioning, quality of life, and medication adherence are assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or schizoaffective disorder
* HAM-D score of 8 or above
* Antipsychotic medication treatment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2001-09; Primary Completion 2006-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sidney Zisook, MD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - San Diego VA Medical Center, San Diego, California
  - Veterans Administration Hospital of Cincinnati, Cincinnati, Ohio

REFERENCES:
- [Derived] Zisook S, Kasckow JW, Lanouette NM, Golshan S, Fellows I, Vahia I, Mohamed S, Rao S. Augmentation with citalopram for suicidal ideation in middle-aged and older outpatients with schizophrenia and schizoaffective disorder who have subthreshold depressive symptoms: a randomized controlled trial. J Clin Psychiatry. 2010 Jul;71(7):915-22. doi: 10.4088/JCP.09m05699gre. Epub 2010 Mar 9. PMID 20361918
- [Derived] Zisook S, Kasckow JW, Golshan S, Fellows I, Solorzano E, Lehman D, Mohamed S, Jeste DV. Citalopram augmentation for subsyndromal symptoms of depression in middle-aged and older outpatients with schizophrenia and schizoaffective disorder: a randomized controlled trial. J Clin Psychiatry. 2009 Apr;70(4):562-71. doi: 10.4088/jcp.08m04261. Epub 2008 Dec 16. PMID 19192468